CLINICAL TRIAL: NCT03631134
Title: Effect of SGLT2 Inhibitor on Blood Glucose Profile in Type 2 Diabetic Patients Using Basal
Brief Title: Effect of SGLT2 Inhibitor on Blood Glucose Profile in Type 2 Diabetic Patients Using Basal Insulin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20170904-02
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SGLT2i treatment (Experimental): The patients who are using basal insulin therapy with or without oral hypoglycemic drugs will be added SGLT2 inhibitor treatment
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Patients will be gave SGLT2 inhibitor 10mg per day

SUMMARY:
The change of glycemic variation and insulin dose after adding SGLT2 inhibitor in type 2 diabetic patients treated with basal insulin was observed in a single center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM, which was defined bypublished Criteria of World Health Organization in 1999;
2. Patients were using glargine with or without oral hypoglycemic drugs and having a stable dose of glargine for more than 2 month would be recruited into this study;
3. Patients had relatively constant diet and exercise in 2 month before the study.
4. Fasting blood glucose was between 6.1 and 16mmolL, and postprandial (or random) blood glucose <22.2mmol/L

Exclusion Criteria:

1. Patients with severe cardiovascular diseases, such as stroke, transient ischemic attack, myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous coronary intervention, and heart failure;
2. Patients with severe infectious diseases;
3. Patients with acute complications of diabetes on admission, such as diabetic ketoacidosis, diabetic hyperosmolar nonketotic coma, and lactic acidosis;
4. Patients with history of psychiatric disorders and were unsuitable to use CGMS;
5. Patients used GLP-1 analogues，SGLT2 or more than once insulin injection in the past 3 months
6. Any other situations that made patients unsuitable to participate in the study, such as alcoholism and drug abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-15 (Estimated); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Changes of glycemic variation | Week 1-5
  Changes of glycemic variation assessed by CGM before and after SGLT2 inhibitor adding

SECONDARY OUTCOMES:
Change of insulin dose | Week 1-5
  Change of insulin dose before and after SGLT2 inhibitor adding